CLINICAL TRIAL: NCT05224271
Title: Patient Reported Outcomes in Radiation Therapy (PRO-RT)
Brief Title: Evaluating Patient Reported Outcomes in Radiation Therapy, the PRO-RT Study
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: ROR2103; NCI-2021-12580 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-003294 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Carcinoma; Head and Neck Carcinoma; Lung Carcinoma; Malignant Solid Neoplasm
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (surveys, medical records & Fitbit collection): Patients complete surveys via the Hugo Platform at baseline (before treatment), after treatment, and at 3 and 6 months after treatment. Patients' medical records and Fitbit information are also collected into the Hugo Platform.
  Interventions: Other: Electronic Health Record Review; Other: Medical Device Usage and Evaluation; Other: Survey Administration

INTERVENTIONS:
Other: Electronic Health Record Review — Medical records are collected
Other: Medical Device Usage and Evaluation — Fitbit information is collected
Other: Survey Administration — Complete surveys

SUMMARY:
This study explores the use of the Hugo platform to involve study participants in their healthcare and treatments. The Hugo platform may allow researchers to collect better and more accurate real-time health data, from other clinics/hospitals, pharmacies and other electronic devices. The purpose of this research is to see if the use of the Hugo platform is consistent, accurate, cost effective, and time efficient, as it collects and transmits important real-time health information from other clinics/hospitals, pharmacies, and other electronic devices.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the data aggregation from a patient centered platform over a follow up period for completeness and quality, including externally linked electronic health record (EHR) information, toxicity completion, and the patient reported outcomes (PRO) response rates for study patients, compared with historical pre-coronavirus disease (COVID) cohort of registry patients.

II. To explore biometric information obtained from wearables as it pertains to the toxicity of treatment for patients using a wearable device.

III. To estimate app-based survey completion rates using Hugo-based survey incentive completion (gift cards).

IV. To explore the cost data available on the platform.

OUTLINE:

Patients complete surveys via the Hugo Platform at baseline (before treatment), after treatment, and at 3 and 6 months after treatment. Patients' medical records and Fitbit information are also collected into the Hugo Platform.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* English speaking
* Consented for Outcomes Registry Study (15-000136)
* Undergoing radiotherapy for cancer treatment with curative intent
* Willing to and able to give consent and participate in study
* Willing to complete all surveys
* Able to access a device (computer, smartphone, or tablet) with web access every day to complete study surveys
* Willing to connect to a device (i.e., a smartphone, Fitbit, or tablet) that can regularly link to Hugo for data transfer
* Willing to share personal information to Tremendous to be able to obtain the Visa e-cards for time and effort put into this study
* Willing to use the Hugo health data sharing platform
* Willing to create a Mayo Clinic Patient Portal (if not already created)

Exclusion Criteria:

* Unable to give consent and enroll prior to administration of baseline survey
* Partial breast radiation therapy (RT) (3 fraction), due to overlap in cadence used for all disease sites
* Stereotactic body radiation therapy (SBRT) to the lung, due to overlap in cadence used for all disease sites
* Co-enrollment on another PRO related study (soft rule)

  * Coordinator would need to get source data from Adam via Hugo
  * Response data will only be accessible by select people

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast, head and neck, and lung tumor types, who are undergoing simulation for treatment in the Radiation Oncology Department at Mayo Clinic
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Survey completion rate | Baseline up to 6 months after completion of radiation therapy
  The difference in rates will be estimated. A chi square, or Fisher's exact test as appropriate, will be used to compare the rates between cohorts. A logistic regression model will be used to understand the association of patient and disease variables with the odds of completion (at least one of the surveys at the treated site).
Percentage of patients with access to wearable device | Up to 6 months after completion of radiation therapy
  A logistic regression model will be used to understand the association of patient and disease variables with the odds of access to a wearable device.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 6 months after completion of radiation therapy
  Logistic regression will be used to predict presence of a patient toxicity. Baseline patient and disease characteristics, along with biometric information will be used to assess associations with toxicity. Multiple variable models will be considered depending on the number of patients identified with a toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly S. Corbin, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials